CLINICAL TRIAL: NCT05000008
Title: Aerobic Versus Anaerobic Exercise on Immune Functions and Disease Severity in Patients With COVID-19: A Randomized Control Trial
Brief Title: Aerobic Versus Anaerobic Exercise on Immune Functions and Disease Severity in Patients With COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Principal Investigator, Motaz Alawna, Assistant Professor, Istanbul Gelisim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Arab American University
Record Dates: First submitted 2021-08-06; First posted 2021-08-11 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Covid19; Immune Response
MeSH Terms: conditions — COVID-19 | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Group (Experimental): Moderate Intensity Aerobic Exercises
  Interventions: Other: Exercises
- Resistance Exercise Group (Experimental): Moderate Intensity Resistance Exercises
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — Moderate aerobic and resistance exercise programe

SUMMARY:
Participants were assigned randomly into two groups, aerobic exercise and resistance exercise groups. All participants in both groups followed the WHO guidelines of quarantine and used standardized medications given by the physician according to the Turkish Ministry of Health guidelines, including the Hydroxyclorocin Sulphate 200 Mg Film Tablet (Plaquenil 200 Mg Film Tablet). The dose was 2 times/ day, 200Mg/time, for 5 days. Besides, the aerobic exercise group performed moderate-intensity aerobic exercises for 40 min/ 3 sessions/week, 40 minute/session, and the resistance exercise groups 40 min/ 3 sessions/week, 40 minute/session.

DETAILED DESCRIPTION:
Evaluative procedures There were two main dependent variables including blood immune markers and severity of respiratory symptoms. These measurements were collected at the baseline after one week and 24 h after the end of the exercise program (two weeks).

A lab technician was asked to visit the patient at home (quarantine). The lab technician wore special protective equipment recommended by WHO. Two visits were performed, one at the beginning of the research procedures, and the last visit at the 24 hours after the end of the exercise program (two weeks). The technician collected blood and saliva samples to be analyzed.

Blood sample collection Blood samples were taken in the morning (8:30-9:30). 10mL of venous blood was collected. Participants were asked to stop any exercise for at least 24 hours before blood sampling. Also, participants were asked to stop eating any food or liquid from 22:00 the prior day of measurement. Samples were collected in vacutainer tubes with sodium ethylenediaminetetraacetic acid (EDTA) for plasma separation. The blood was centrifuged at 3,000 rpm for 15 min at 4◦C. The investigators measured total lymphocytes, leukocytes, and monocytes from total-blood samples utilizing a multichannel hemocyte analysis system (SE-9000; Sysmex Corp, Hyogo, Japan). The concentrations of IL-6, IL-10, and TNF-α were analyzed by using ELISA commercial kits assay (R&D Systems, Minneapolis, USA) following the manufacturer's instructions for analysis on an EZ-Reader microplate reader at 450 nm. The samples were stored at -20◦C for further analysis.

Saliva sample collection A saliva sample was collected to measure the salivary IgA-S concentration. The saliva sample was taken without any saliva stimulation methods, the participant was asked to rinse their mouths with distilled water and to evacuate their mouth just before collection. The investigators used the passive drainage method for the collection, in which the participant slightly flexed their head forward to allow the saliva to move into a sterilized and pre-weighed Falcon tube for 5min. The weight of tubes were measured again following collection, to estimate the volume and the saliva flow rate. The tubes were weighed with 0.1mg accuracy with proposed saliva density as 1.0 g.mL-1. The samples were stored at -80◦C for further analysis. The S-IgA concentration were analyzed utilizing commercial ELISA kits (IgA Salivary, DRG, Minneapolis, USA). The IgA-S secretion rate (ng/min) was measured by multiplying the whole concentration of IgA-S present in the mucosal surface per unit of time by the saliva flow rate (mL/min).

Wisconsin Upper Respiratory Symptom Survey the Wisconsin Upper Respiratory Symptom Survey (WURSS) is an empirically derived patient-oriented illness-specific quality-of-life evaluative outcomes instrument. The development process of this survey was described in detail by Barrett et al. WURSS-24 is designed to evaluate the negative effect of acute upper respiratory infection, presumed viral (the common cold). It is a valid and reliable measurement tool to evaluate the measure items and domains that change over time including influenza-like illness symptoms of headache, body aches, and fever. The participants were asked to fill the survey before starting the study and the 2 times/week.

Treatment Procedures Participants were assigned randomly into two groups, exercise and control groups. All participants in both groups followed the WHO guidelines of quarantine and used standardized medications given by the physician according to the Turkish Ministry of Health, including the Hydroxyclorocin Sulphate 200 Mg Film Tablet (Plaquenil 200 Mg Film Tablet). The dose was 2 times/ day, 200Mg/time, for 5 days Besides, the exercise group performed a moderate-intensity aerobic exercises for 40 min/ 3 sessions/week, 40 minute/session.

Participants in the aerobic exercise group performed a two weeks aerobic exercise program. The exercise program consisted of walking/running on a treadmill or bicycling on a stationary bicycle. Each session is composed of five-minute warm-up slow walking or bicycling. Then the main intervention which composed of thirty-minutes of moderate-intensity aerobic exercises (walking/running or bicycling). Lastly, a five-minute of cool-down exercise (walking/running or bicycling). The exercise intensity was 60-75% of the predicted MHR (calculated as MHR=210-age).

The resistance exercises program consists of 3 sessions/week, 60 min/session for 2 weeks. The two-way body part split protocol was used during the resistance exercises (legs, back and biceps on one day; chest, shoulders and triceps on a separate day) alternatively. During each session group of 5 exercises have been performed using both multi-joint and single joint exercises. A 5 - 10 min of warm up exercises have been before the beginning of each session, warm up exercises consist of moderate speed walking and stretching exercises. Three set of exercises have been performed with 1 - 2 min rest between sets. During the first week the resistance exercises intensity has been adjusted to be eight repetitions for each exercise at 70% of 1RM, During the second week, the intensity was increased to 80% of 1 RM.

The Borg Rating of Perceived Exertion (RPE) scale was used to control the exercise intensity. PRE is a reliable and validated scale to allow individuals to monitor and guide the exercise intensity by rating their level of exertion during exercise. After explaining the scale in detail for the patients, investigators asked them to keep the exertion rating level between 12 to 14 (light - somewhat hard) on the Borg Scale, which suggests that the patient is exercising on a moderate exercise level. The exercise was stopped if the patients experienced any of the following signs and symptoms: chest pain, shortness of breath, fainting, claudication, fatigue, ataxia, dizziness, cyanosis, or pallor.

ELIGIBILITY:
Inclusion Criteria:

* the patient has a recent mild or moderate COVID-19 with no or low-grade fever 99.5- 100.94 °F (37.5-38.3 °C). Mild COVID-19 included that the patient has symptoms of acute upper respiratory tract infection (fever, cough, myalgia, runny nose, fatigue, sore throat, sneezing) or gastrointestinal symptoms (nausea, vomiting, abdominal pain, diarrhea). Moderate grade of COVID 19 included that the participant has pneumonia (cough, frequent fever) with no obvious hypoxemia, the presence of lesions on chest CT

Exclusion Criteria:

* that patient was not hospitalized and has moderate or high-grade fever <100.94 °F (<38.3 °C) or other chronic diseases such as heart problems, hypertension or diabetes. Women how were using contraceptives were excluded due to contraceptives decrease immune functions and might affect the subjectivity to autoimmune disorders with marked increases in risk for various autoimmune disorders

Ages: 24 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Immune Biomarkers | 10 Months
  Blood sample collection,Saliva sample collection,Wisconsin Upper Respiratory Symptom Survey

CONTACTS AND LOCATIONS:
Locations (1):
- Motaz Alawna, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No